CLINICAL TRIAL: NCT00076505
Title: Bioenergetic Function in Parkinson's Disease
Brief Title: Cell Studies of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040092; 04-HG-0092
Record Dates: First submitted 2004-01-23; First posted 2004-01-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-11-30

CONDITIONS: Parkinson Disease
Keywords: Mitochondria; Proteasome; Lipid; Polymorphism; Genetic; Parkinson's Disease; Parkinson Disease; PD; Heredity; Parkinson Disease At Risk; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
This study will examine and compare blood samples from healthy volunteers and patients with Parkinson's disease to identify abnormalities associated with Parkinson's disease. Disease symptoms include slowness of movement, hand or leg shaking, and stiffness. Some patients have difficulty with balance. Information from this study may provide information on how Parkinson's disease affects the brain and body, and may help lead to a test for earlier diagnosis.

Healthy volunteers and patients with Parkinson's disease who are 18 years of age or older may enroll in this study. Participants will undergo the following procedures:

* Physical examination, including evaluation of strength, feeling, coordination, and balance
* Blood drawing: 150 milliliters (about 10 tablespoons) of blood will be drawn
* Personal and family medical history
* Consent to access medical records for research purposes

Blood samples will be examined for:

* Genetic analysis
* Study of specific proteins and lipids
* Study of mitochondria (parts of cells that make energy)

DETAILED DESCRIPTION:
This study wants to focus on mitochondrial defects associated with Parkinson's disease (PD) and how they relate to alpha-synuclein (SNCA) expression and function. Individuals from families with inherited Parkinson's disease (affected and at risk members), as well as normal individuals, will be enrolled. All subjects will be asked to provide blood samples in order to study bioenergetic function in mitochondria from their platelets. These studies will include genotyping and determination of polymorphisms in the subjects' mitochondrial DNA (mtDNA) in order to delineate any significant abnormality that may be associated with a particular group. Cardiolipin levels will be obtained fee for service at Lipomics. Basic respirometry, enzyme activity, and somatic cell hybridization will be performed in the PI's lab. Protein analysis will be performed in the proteomics facility at NIMH.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals over the age of 18 from families in which an inherited form of parkinson's disease is apparent will be enrolled. These patients are already enrolled in the Genetic linkage analysis protocol 97-HG-0173.

The diagnosis of Parkinson's disease must be supported by accepted clinical criteria including: tremor, bradykinesia, rigidity and responsiveness to L-DOPA.

Unaffected family members found to be at risk, will also be enrolled.

The normal control group will be comprised of anonymous platelet donors from the NIH Department of Transfusion Medicine and of individuals over the age of 18 with no known neurological disorder and normal neurological examination matched by age and sex that may be actively recruited.

Individuals with Lewy Body disease (LBD) that meet current criteria for diagnosis (hallucinations, diurnal variation, and dementia associated with extrapyramidal symptoms within a one year period) will also be included in the study.

EXCLUSION CRITERIA:

Because some medications can alter mitochondrial function, patients on MAO inhibitors, antidiabetic sulfonylureas and benzodiazepines will be excluded from the study.

No person under the age of 18 will be enrolled in this study. This is due to the fact that, except for very rare occasions, Parkinson's disease affects only adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-01-14; Study Completion 2006-11-30

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Leroy E, Boyer R, Auburger G, Leube B, Ulm G, Mezey E, Harta G, Brownstein MJ, Jonnalagada S, Chernova T, Dehejia A, Lavedan C, Gasser T, Steinbach PJ, Wilkinson KD, Polymeropoulos MH. The ubiquitin pathway in Parkinson's disease. Nature. 1998 Oct 1;395(6701):451-2. doi: 10.1038/26652. No abstract available. PMID 9774100